CLINICAL TRIAL: NCT05651256
Title: Preliminary Findings of the Efficacy of Botulinum Toxin in Temporomandibular Disorders: A Randomized Clinical Trial
Brief Title: Efficacy of Botulinum Toxin in Temporomandibular Disorders
Acronym: TMD
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, JAVIER MONTERO, Professor, University of Salamanca
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PI 2021 04 734
Record Dates: First submitted 2022-11-15; First posted 2022-12-14 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Temporomandibular Joint Disorder Bilateral
Keywords: Botulinum toxin; Temporomandibular joint disorders; Masticatory disfunction syndrome; Randomized clinical trial
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TREATMENT (Experimental): BEFORE TREATMENT/AFTER TREATMENT A 1 cc marked insulin syringe was used for intramuscular injection of the prepared solution, according to the locations and amounts proposed with a total dose of 100 U (Type A toxinum botulinum, Allergan) in each patient, distributed at the different injection sites: 40 U in the masseter muscle, (0.1 cc=10 U), 20 U in the area of greatest hypertrophy (anterior inferior masseter), 10 U in the direction of the mandibular inferior border and 10 U in the area of the posterior inferior masseter; 20 U in the lateral pterygoid muscle (10 U extraorally between the zygomatic arch and sigmoid notch and 10 U intraorally, behind the maxillary tuberosity); 20 U in the TMJ, 10mm anterior to the tragus and 2mm below the zygomatic arch and 20 U in the anterior part of the temporalis muscle.
  Interventions: Drug: Botulinum toxin type A injection

INTERVENTIONS:
Drug: Botulinum toxin type A injection — The solution for injection was prepared immediately before the intervention, by dissolving the vials of BTX, kept refrigerated at 5ºC, in 1 ml of sterile saline solution at room temperature. Eight injection sites were marked, three located in the masseter muscle, two in the lateral pterygoid muscle, one in the temporomandibular joint (TMJ) and two in the temporalis muscle. A 1 cc marked insulin syringe was used for intramuscular injection of the prepared solution, according to the locations and amounts proposed by Kim et al. and Ho et al. with a total dose of 100 U in each patient.distributed at the different injection sites.
  Other Names: Botox® 100 U, Allergan Pharmaceuticals Westport, Ireland

SUMMARY:
Temporomandibular disorders (TMDs) represent a multifactorial pathological group that gives rise to a varied and complex symptomatology that includes decreased jaw movement, muscle and joint pain, joint crepitation and limitation or functional deviation of the jaw opening.

All this is sometimes accompanied by headache and other painful symptoms in the neck musculature, incapacitating for many patients and at considerable public health expense. Intramuscular and intra-articular injections of botulinum toxin are a simple treatment that has proven to be effective in the treatment of the painful symptoms of these disorders, being a therapeutic option in situations of failure of conventional treatments, without presenting adverse effects.

Our study presents the preliminary results of twenty patients treated with this therapy

DETAILED DESCRIPTION:
TMDs are a common pathology affecting up to 70% of the population, with a maximum incidence in young patients. We used a sample of twenty patients recruited in the Maxillofacial Surgery Service of the University Hospital of Salamanca (Spain), who met the inclusion criteria, with unilateral painful symptomatology of more than three months duration. All patients were randomly treated by intramuscular and intra-articular injections of BTX (100 U) in 8 predetermined points. Pain symptomatology was assessed at the different locations, together with joint symptomatology, at baseline and 6 weeks after treatment.

Adverse effects were also evaluated. In 85% of the patients, pain on oral opening improved and 90% showed improvement of pain on mastication. A 75% of the patients reported improvement in joint clicking/noise. Headaches improved or disappeared in 70% of the patients treated. Despite the limitations of the study and the preliminary results, intramuscular and intra-articular infiltrations with BTX were effective in the treatment of symptoms associated with TMDs, with minimal adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* The study included patients diagnosed with TMDs, according to the established diagnostic criteria, aged between 18 and 69 years (both included) and with unilateral painful symptomatology of more than three months' duration.

Exclusion Criteria:

* Patients previously treated with surgery/arthrocentesis of the TMJ; patients treated in the last six months with surgery in the cervicofacial region; patients who, at the time of inclusion in the study, were being treated in a "Pain Unit" and patients who had previously received treatment with BTX.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Measurement of pain intensity in the masticatory musculature | 6 weeks
  Pain intensity was evaluated through the visual analogue scale (VAS). The patients determined the intensity of pain in the different locations of the craniofacial region (temporal muscle, masseter muscle, pterygoid muscle, and TMJ) in a range of 0 to 10, before and after the administration of botulinum toxin.
  0 was the absence of pain and 10 the intensity of maximum pain. The percentage of patients in whom the pain intensity of the masticatory muscles decreased after treatment with botox type A was analyzed.
Complications in the administration of botulinum toxin | 6 weeks
  Adverse side effects assessed included warmth, redness, and bruising at the injection site, swallowing disturbance, contracture or pain of the contralateral muscle, and abnormal jaw movements.
  Therefore, the percentage of patients included in the study who presented complications after the injection of botulinum toxin according to the established parameters was analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: JAVIER MONTERO, PROFESSOR, Study Director — Salamanca University
Locations (1):
- Clinica Odontológica de la Universidad de Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schiffman E, Ohrbach R, Truelove E, Look J, Anderson G, Goulet JP, List T, Svensson P, Gonzalez Y, Lobbezoo F, Michelotti A, Brooks SL, Ceusters W, Drangsholt M, Ettlin D, Gaul C, Goldberg LJ, Haythornthwaite JA, Hollender L, Jensen R, John MT, De Laat A, de Leeuw R, Maixner W, van der Meulen M, Murray GM, Nixdorf DR, Palla S, Petersson A, Pionchon P, Smith B, Visscher CM, Zakrzewska J, Dworkin SF; International RDC/TMD Consortium Network, International association for Dental Research; Orofacial Pain Special Interest Group, International Association for the Study of Pain. Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) for Clinical and Research Applications: recommendations of the International RDC/TMD Consortium Network* and Orofacial Pain Special Interest Groupdagger. J Oral Facial Pain Headache. 2014 Winter;28(1):6-27. doi: 10.11607/jop.1151. PMID 24482784
- [Background] Okeson JP. Current terminology and diagnostic classification schemes. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 1997 Jan;83(1):61-4. doi: 10.1016/s1079-2104(97)90092-5. PMID 9007925
- [Background] Liu F, Steinkeler A. Epidemiology, diagnosis, and treatment of temporomandibular disorders. Dent Clin North Am. 2013 Jul;57(3):465-79. doi: 10.1016/j.cden.2013.04.006. PMID 23809304
- [Background] Kobayashi FY, Gaviao MB, Montes AB, Marquezin MC, Castelo PM. Evaluation of oro-facial function in young subjects with temporomandibular disorders. J Oral Rehabil. 2014 Jul;41(7):496-506. doi: 10.1111/joor.12163. Epub 2014 Mar 24. PMID 24661101
- [Background] Baba K, Tsukiyama Y, Yamazaki M, Clark GT. A review of temporomandibular disorder diagnostic techniques. J Prosthet Dent. 2001 Aug;86(2):184-94. doi: 10.1067/mpr.2001.116231. PMID 11514808
- [Background] Gauer RL, Semidey MJ. Diagnosis and treatment of temporomandibular disorders. Am Fam Physician. 2015 Mar 15;91(6):378-86. PMID 25822556
- [Background] Lomas J, Gurgenci T, Jackson C, Campbell D. Temporomandibular dysfunction. Aust J Gen Pract. 2018 Apr;47(4):212-215. doi: 10.31128/AFP-10-17-4375. PMID 29621862
- [Background] Shoohanizad E, Garajei A, Enamzadeh A, Yari A. Nonsurgical management of temporomandibular joint autoimmune disorders. AIMS Public Health. 2019 Dec 12;6(4):554-567. doi: 10.3934/publichealth.2019.4.554. eCollection 2019. PMID 31909075
- [Background] Ta LE, Dionne RA. Treatment of painful temporomandibular joints with a cyclooxygenase-2 inhibitor: a randomized placebo-controlled comparison of celecoxib to naproxen. Pain. 2004 Sep;111(1-2):13-21. doi: 10.1016/j.pain.2004.04.029. PMID 15327804
- [Background] Herman CR, Schiffman EL, Look JO, Rindal DB. The effectiveness of adding pharmacologic treatment with clonazepam or cyclobenzaprine to patient education and self-care for the treatment of jaw pain upon awakening: a randomized clinical trial. J Orofac Pain. 2002 Winter;16(1):64-70. PMID 11889661
- [Background] Hersh EV, Balasubramaniam R, Pinto A. Pharmacologic management of temporomandibular disorders. Oral Maxillofac Surg Clin North Am. 2008 May;20(2):197-210, vi. doi: 10.1016/j.coms.2007.12.005. PMID 18343325
- [Background] Park J, Park HJ. Botulinum Toxin for the Treatment of Neuropathic Pain. Toxins (Basel). 2017 Aug 24;9(9):260. doi: 10.3390/toxins9090260. PMID 28837075
- [Background] Fallah HM, Currimbhoy S. Use of botulinum toxin A for treatment of myofascial pain and dysfunction. J Oral Maxillofac Surg. 2012 May;70(5):1243-5. doi: 10.1016/j.joms.2012.01.015. No abstract available. PMID 22538024
- [Background] Patel J, Cardoso JA, Mehta S. A systematic review of botulinum toxin in the management of patients with temporomandibular disorders and bruxism. Br Dent J. 2019 May;226(9):667-672. doi: 10.1038/s41415-019-0257-z. PMID 31076698
- [Background] Serrera-Figallo MA, Ruiz-de-Leon-Hernandez G, Torres-Lagares D, Castro-Araya A, Torres-Ferrerosa O, Hernandez-Pacheco E, Gutierrez-Perez JL. Use of Botulinum Toxin in Orofacial Clinical Practice. Toxins (Basel). 2020 Feb 11;12(2):112. doi: 10.3390/toxins12020112. PMID 32053883
- [Background] von Lindern JJ, Niederhagen B, Berge S, Appel T. Type A botulinum toxin in the treatment of chronic facial pain associated with masticatory hyperactivity. J Oral Maxillofac Surg. 2003 Jul;61(7):774-8. doi: 10.1016/s0278-2391(03)00153-8. PMID 12856249
- [Background] Munoz Lora VRM, Del Bel Cury AA, Jabbari B, Lackovic Z. Botulinum Toxin Type A in Dental Medicine. J Dent Res. 2019 Dec;98(13):1450-1457. doi: 10.1177/0022034519875053. Epub 2019 Sep 18. PMID 31533008
- [Background] Kim NH, Park RH, Park JB. Botulinum toxin type A for the treatment of hypertrophy of the masseter muscle. Plast Reconstr Surg. 2010 Jun;125(6):1693-1705. doi: 10.1097/PRS.0b013e3181d0ad03. PMID 20517093
- [Background] Ho KY, Tan KH. Botulinum toxin A for myofascial trigger point injection: a qualitative systematic review. Eur J Pain. 2007 Jul;11(5):519-27. doi: 10.1016/j.ejpain.2006.09.002. Epub 2006 Oct 27. PMID 17071119
- [Background] Sidebottom AJ, Patel AA, Amin J. Botulinum injection for the management of myofascial pain in the masticatory muscles. A prospective outcome study. Br J Oral Maxillofac Surg. 2013 Apr;51(3):199-205. doi: 10.1016/j.bjoms.2012.07.002. Epub 2012 Aug 4. PMID 22871559
- [Background] Laskin DM. The Use of Botulinum Toxin for the Treatment of Myofascial Pain in the Masticatory Muscles. Oral Maxillofac Surg Clin North Am. 2018 Aug;30(3):287-289. doi: 10.1016/j.coms.2018.04.004. Epub 2018 Jul 5. PMID 30008341
- [Background] Soares A, Andriolo RB, Atallah AN, da Silva EM. Botulinum toxin for myofascial pain syndromes in adults. Cochrane Database Syst Rev. 2014 Jul 25;2014(7):CD007533. doi: 10.1002/14651858.CD007533.pub3. PMID 25062018
- [Background] Freund B, Schwartz M, Symington JM. The use of botulinum toxin for the treatment of temporomandibular disorders: preliminary findings. J Oral Maxillofac Surg. 1999 Aug;57(8):916-20; discussion 920-1. doi: 10.1016/s0278-2391(99)90007-1. PMID 10437718
- [Background] Freund B, Schwartz M, Symington JM. Botulinum toxin: new treatment for temporomandibular disorders. Br J Oral Maxillofac Surg. 2000 Oct;38(5):466-71. doi: 10.1054/bjom.1999.0238. PMID 11010775
- [Background] Nayyar P, Kumar P, Nayyar PV, Singh A. BOTOX: Broadening the Horizon of Dentistry. J Clin Diagn Res. 2014 Dec;8(12):ZE25-9. doi: 10.7860/JCDR/2014/11624.5341. Epub 2014 Dec 5. PMID 25654058
- [Background] Hoque A, McAndrew M. Use of botulinum toxin in dentistry. N Y State Dent J. 2009 Nov;75(6):52-5. PMID 20069790
- [Background] Al-Wayli H. Treatment of chronic pain associated with nocturnal bruxism with botulinum toxin. A prospective and randomized clinical study. J Clin Exp Dent. 2017 Jan 1;9(1):e112-e117. doi: 10.4317/jced.53084. eCollection 2017 Jan. PMID 28149474
- [Background] Satriyasa BK. Botulinum toxin (Botox) A for reducing the appearance of facial wrinkles: a literature review of clinical use and pharmacological aspect. Clin Cosmet Investig Dermatol. 2019 Apr 10;12:223-228. doi: 10.2147/CCID.S202919. eCollection 2019. PMID 31114283
- [Background] Srivastava S, Kharbanda S, Pal US, Shah V. Applications of botulinum toxin in dentistry: A comprehensive review. Natl J Maxillofac Surg. 2015 Jul-Dec;6(2):152-9. doi: 10.4103/0975-5950.183860. PMID 27390488
- [Background] Laskin DM. Botulinum toxin A in the treatment of myofascial pain and dysfunction: the case against its use. J Oral Maxillofac Surg. 2012 May;70(5):1240-2. doi: 10.1016/j.joms.2011.05.030. No abstract available. PMID 22538023
- [Background] Pihut M, Ferendiuk E, Szewczyk M, Kasprzyk K, Wieckiewicz M. The efficiency of botulinum toxin type A for the treatment of masseter muscle pain in patients with temporomandibular joint dysfunction and tension-type headache. J Headache Pain. 2016;17:29. doi: 10.1186/s10194-016-0621-1. Epub 2016 Mar 24. PMID 27011213
- [Background] Chikhani L, Dichamp J. [Bruxism, temporo-mandibular dysfunction and botulinum toxin]. Ann Readapt Med Phys. 2003 Jul;46(6):333-7. doi: 10.1016/s0168-6054(03)00115-6. French. PMID 12928140
- [Background] Hosgor H, Altindis S. Efficacy of botulinum toxin in the management of temporomandibular myofascial pain and sleep bruxism. J Korean Assoc Oral Maxillofac Surg. 2020 Oct 31;46(5):335-340. doi: 10.5125/jkaoms.2020.46.5.335. PMID 33122458
- [Background] Patel AA, Lerner MZ, Blitzer A. IncobotulinumtoxinA Injection for Temporomandibular Joint Disorder. Ann Otol Rhinol Laryngol. 2017 Apr;126(4):328-333. doi: 10.1177/0003489417693013. Epub 2017 Feb 1. PMID 28290229
- [Background] Thomas NJ, Aronovich S. Does Adjunctive Botulinum Toxin A Reduce Pain Scores When Combined With Temporomandibular Joint Arthroscopy for the Treatment of Concomitant Temporomandibular Joint Arthralgia and Myofascial Pain? J Oral Maxillofac Surg. 2017 Dec;75(12):2521-2528. doi: 10.1016/j.joms.2017.04.011. Epub 2017 Apr 19. PMID 28500876
- [Background] Batifol D. [Different types of injection in temporomandibular disorders (TMD) treatment]. Rev Stomatol Chir Maxillofac Chir Orale. 2016 Sep;117(4):256-8. doi: 10.1016/j.revsto.2016.07.005. Epub 2016 Aug 23. French. PMID 27561987
- [Background] Gadhia K, Walmsley D. The therapeutic use of botulinum toxin in cervical and maxillofacial conditions. Evid Based Dent. 2009;10(2):53. doi: 10.1038/sj.ebd.6400654. PMID 19561583
- [Background] Blumenfeld AM, Stark RJ, Freeman MC, Orejudos A, Manack Adams A. Long-term study of the efficacy and safety of OnabotulinumtoxinA for the prevention of chronic migraine: COMPEL study. J Headache Pain. 2018 Feb 5;19(1):13. doi: 10.1186/s10194-018-0840-8. PMID 29404713
- [Background] Binder WJ, Brin MF, Blitzer A, Schoenrock LD, Pogoda JM. Botulinum toxin type A (BOTOX) for treatment of migraine headaches: an open-label study. Otolaryngol Head Neck Surg. 2000 Dec;123(6):669-76. doi: 10.1067/mhn.2000.110960. PMID 11112955
- [Background] Freund BJ, Schwartz M. Treatment of chronic cervical-associated headache with botulinum toxin A: a pilot study. Headache. 2000 Mar;40(3):231-6. doi: 10.1046/j.1526-4610.2000.00033.x. PMID 10759926
- [Background] Freund BJ, Schwartz M. Treatment of whiplash associated neck pain [corrected] with botulinum toxin-A: a pilot study. J Rheumatol. 2000 Feb;27(2):481-4. PMID 10685817
- [Background] Ihde SK, Konstantinovic VS. The therapeutic use of botulinum toxin in cervical and maxillofacial conditions: an evidence-based review. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2007 Aug;104(2):e1-11. doi: 10.1016/j.tripleo.2007.02.004. Epub 2007 Jun 7. PMID 17560141
- [Background] Blitzer A, Sulica L. Botulinum toxin: basic science and clinical uses in otolaryngology. Laryngoscope. 2001 Feb;111(2):218-26. doi: 10.1097/00005537-200102000-00006. PMID 11210864
- [Background] Sari BC, Develi T. The effect of intraarticular botulinum toxin-A injection on symptoms of temporomandibular joint disorder. J Stomatol Oral Maxillofac Surg. 2022 Oct;123(5):e316-e320. doi: 10.1016/j.jormas.2022.04.019. Epub 2022 May 14. PMID 35523405
- [Background] Lora VR, Clemente-Napimoga JT, Abdalla HB, Macedo CG, Canales GT, Barbosa CM. Botulinum toxin type A reduces inflammatory hypernociception induced by arthritis in the temporomadibular joint of rats. Toxicon. 2017 Apr;129:52-57. doi: 10.1016/j.toxicon.2017.02.010. Epub 2017 Feb 14. PMID 28209481
- [Background] Drinovac Vlah V, Filipovic B, Bach-Rojecky L, Lackovic Z. Role of central versus peripheral opioid system in antinociceptive and anti-inflammatory effect of botulinum toxin type A in trigeminal region. Eur J Pain. 2018 Mar;22(3):583-591. doi: 10.1002/ejp.1146. Epub 2017 Nov 13. PMID 29134730
- [Background] Sipahi Calis A, Colakoglu Z, Gunbay S. The use of botulinum toxin-a in the treatment of muscular temporomandibular joint disorders. J Stomatol Oral Maxillofac Surg. 2019 Sep;120(4):322-325. doi: 10.1016/j.jormas.2019.02.015. Epub 2019 Feb 23. PMID 30807862
- [Derived] Macedo de Sousa B, Lopez-Valverde N, Ferreira C, de Almeida AM, Lopez-Valverde A, Blanco Rueda JA. Efficacy of botulinum toxin type A in myogenic temporomandibulardisorders: a single arm, prospective, pilot study. Front Rehabil Sci. 2025 Dec 19;6:1737706. doi: 10.3389/fresc.2025.1737706. eCollection 2025. PMID 41487935